CLINICAL TRIAL: NCT00496665
Title: A Phase I Study of ZD6474 (Zactima) and Metronomic Chemotherapy in Advanced Breast Cancer
Brief Title: ZD6474 (Zactima) and Metronomic Chemotherapy in Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AstraZeneca (Industry); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Erica Mayer, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-402
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Stage IV breast cancer; metronomic chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — vandetanib; Cyclophosphamide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vandetenib (Experimental): Cyclophosphamide 50 mg daily, methotrexate 2.5 mg days 1-2 weekly, and daily vandetanib (zactima) in 3 dose-escalation cohorts (100mg=Cohort 1) (200mg=Cohort 2) (300mg=Cohort3)
  Interventions: Drug: Vandetanib; Drug: Cyclophosphamide; Drug: Methotrexate

INTERVENTIONS:
Drug: Vandetanib — Taken orally once a day in 28-day cycles (the dose will vary)
  Other Names: Zactima; ZD6474
Drug: Cyclophosphamide — Metronic Chemotherapy: Low dose pills taken every day of each 28-day cycle
Drug: Methotrexate — Metronic Chemotherapy: low dose pills taken on days 1 and 2 of each week

SUMMARY:
The purpose of this research study is to determine the safety and tolerability of the combination of Zactima with metronomic chemotherapy. Zactima is an oral anti-angiogenesis drug, which means it fights cancer by cutting off a tumor's blood supply. Thus, the drug starves the tumor by preventing the delivery of nutrients and oxygen. Metronomic chemotherapy is low dose oral chemotherapy pills which are taken daily. Unlike traditional chemotherapy, metronomic chemotherapy is thought to fight cancer like Zactima, by cutting off the blood supply to tumors. Because the dose is very low, the side effects are generally mild and very different from those with higher dose chemotherapy given by vein.

DETAILED DESCRIPTION:
* Each study cycle is 28 days long. Participants will take the study drug, Zactima, by mouth once a day. The dose of Zactima the participant will receive will be determined by the time when they enroll on the study. They will also take the metronomic chemotherapy by mouth. This consists of two drugs: cyclophosphamide and methotrexate. Cyclophosphamide is taken every day and methotrexate is taken on days 1 and 2 of each week.
* A physical exam will be performed on Day 1 of each cycle. Vital signs, including height, weight, blood pressure, and temperature will be done on Day 1 of each cycle, as well as at week 3 of Cycles 1 and 2.
* Electrocardiograms will be performed at various points to assess heart function. This will be done at week 1, 3, 5, 7, and 9, and then every 3 months for the rest of the study.
* Routine blood tests will be done on Day 1 of each cycle, as well as at week 3 for the first two cycles. Urine tests will be done on Day 1 of each cycle.
* An ultrasound will be done at Brigham and Women's Hospital in the Department of Vascular Medicine at week 3 and week 7.
* Participants will have scans done to assess their tumor every 2 cycles (8 weeks). These may include a CT scan, MRI, PET scan, x-rays, and/or bone scans.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed Stage IV breast cancer
* Patients may have prior treatment with 0-4 prior chemotherapeutic regimens for metastatic disease.
* 18 years of age and older
* Life expectancy of greater than 3 months as assessed by patient's primary oncologist
* ECOG Performance Status of 0-2.
* LVEF > 45%, as assessed by echocardiogram or nuclear medicine gate study within 30 days prior to initiating protocol-based treatment
* Negative Serum pregnancy test
* No receipt of any investigational agents within 30 days prior to commencing study treatment

Exclusion Criteria:

* Abnormal laboratory results as outlined in the protocol
* Therapeutic anti-coagulation. The use of low dose warfarin, intermittent doses of TPA, or heparin flushes to prophylax against central venous catheter associated clots is acceptable.
* Brain metastases or spinal cord compression, unless treated at least 4 weeks before entry and stable without steroid treatment for one week. Leptomeningeal disease is not eligible.
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate
* Clinically significant cardiac event such as myocardial infarction; NYHA classification of heart disease greater than or equal to 2; or presence of cardiac disease that increases the risk of ventricular arrhythmia
* History of arrhythmia which is symptomatic or requires treatment or asymptomatic sustained ventricular tachycardia
* Previous history of QTc prolongation as a result from other medication that required discontinuation of that medication
* Congenital long QT syndrome, or 1st degree relative with unexplained sudden death under 40 years of age
* Presence of left bundle branch block
* QTc with Bazett's correction that is unmeasurable or greater than 480msec on screening ECG.
* Any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes or induce CYP3A4 function
* Hypertension not controlled by medical therapy
* Currently active diarrhea that may affect the ability of the patient to absorb the Zactima or tolerate diarrhea
* Previous or current non-breast malignancies within the last 5 years, with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy
* Patients with large or rapidly accumulating pleural or abdominal effusions
* Women who are currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of combination therapy with ZD6474 (Zactima) and metronomic chemotherapy | 2 years

SECONDARY OUTCOMES:
To determine the response rate of combination therapy with ZD6474 (Zactima) and metronomic chemotherapy in patients with measurable disease. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Erica Mayer, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts